CLINICAL TRIAL: NCT04103957
Title: Exploring the Effect of Visual Feedback on Motion Trajectory in a Virtual Reality Environment.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201907130RINB
Record Dates: First submitted 2019-09-24; First posted 2019-09-26 (Actual); Last update posted 2021-05-26 (Actual); Status verified 2021-05

CONDITIONS: Stroke; Control
Keywords: Virtual reality
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The rehabilitation intensity and frequency of upper extremities of stroke patients is insufficient. Virtual reality technique may solved this problem. The investigators want to build up the motion trajectory system by head-mounted display virtual reality technique, and to explore the effect of visual feedback on motion trajectory in a virtual reality environment.

DETAILED DESCRIPTION:
How to increase the rehabilitation intensity in the critical rehabilitation window for stroke patients (half year since onset) was very important. The training intensity and frequency of upper extremities is insufficient. The proprioceptive neuromuscular facilitation (PNF) movements of upper extremities are applied to all daily upper extremities movement. The goals of this study are that the investigators want to build up the motion trajectory system by head-mounted display virtual reality technique, and the investigators want to explore the effect of visual feedback on motion trajectory in a virtual reality environment. The investigators will record the motion patterns, motion trajectory and the deviation of position and angle comparing to the normal PNF movement pattern to analyze the motion accuracy.

ELIGIBILITY:
Stroke patients Inclusion criteria

1. Age:20~100y/o.
2. Stroke onset time > 1 week, and neurological status and medical condition are stable.
3. Brunnstrom stage III to V.
4. Can follow order.

Exclusion criteria

1. Crucial organ failure, including heart, lung, liver, and kidney.
2. Brain operation and epilepsy.
3. Severe metal illness and aphasia, so cannot follow order
4. Feel uncomfortable while using virtual reality.
5. Crucial eye problems, including color-blind, weak color, cataract, glaucoma, etc.
6. Mental illness, neuro-musculoskeletal system lesions, vertigo, claustrophobic.
7. Illness and pain to affect upper extremities movement.

Healthy people Inclusion criteria

1. Age:20~100y/o.
2. No pain to affect upper extremities movement.

Exclusion criteria

1. Feel uncomfortable while using virtual reality.
2. Crucial eye problems, including color-blind, weak color, cataract, glaucoma, etc.
3. Cognition impairment, history of mental illness, neuro-musculoskeletal system lesions, vertigo, claustrophobic.
4. Epilepsy.

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Stroke patients Healthy people
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-04-10 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Motion accuracy | during the experiment
  Record the motion patterns, motion trajectory and the deviation of position and angle comparing to the normal PNF movement pattern to analyze the motion accuracy

CONTACTS AND LOCATIONS:
Overall Officials: Tzu Ling Tai, MAMS, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Zhongzheng Dist, Taiwan